CLINICAL TRIAL: NCT03185702
Title: UTHealth Turner Syndrome Research Registry
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Siddharth Prakash, Associate Professor, Internal Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0120
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Saliva, blood, and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Turner Syndrome: Chromosomal diagnosis and typical features
  Interventions: Genetic: Research genetic tests
- Unaffected controls: Normal females and unaffected family members
  Interventions: Genetic: Research genetic tests

INTERVENTIONS:
Genetic: Research genetic tests — DNA and tissue-based tests: karyotype, copy number variants, genome-wide association studies and induced pluripotent stem cells

SUMMARY:
The investigators will conduct genetic comparisons between Turner Syndrome (TS) patients with and without Bicuspid Aortic Valve (BAV) to identify causative agents of BAV in people with TS.

The investigators will correlate the patterns and prevalence of structural heart defects in TS women with emerging molecular data to identify patients who are at high risk for cardiovascular complications

DETAILED DESCRIPTION:
Turner syndrome (TS) is a common chromosomal disorder that affects approximately 1 in 2500 live female births. Complete or partial monosomy of one of the X chromosomes in a female is associated with various congenital heart defects (CHDs), which include aortic dilatation, coarctation of aorta and BAV. Congenital cardiovascular defects related to CHD are the leading cause of death in women with TS. The Turner Syndrome Network Registry (TRN Registry) and genetic sample repository can address gaps in knowledge of CHD in TS by facilitating the recognition of demographic and genetic patterns. TRN Registry-based research can improve surveillance of TS patients who are at risk for CHD and provide valuable insight into genetic components of CHD.

The investigators will recruit TS patients into the TRN Registry and obtain blood and/or saliva samples after informed consent. The genetic diagnosis of TS will be confirmed using chromosomal microarrays. The array data will be also be used to identify genomic copy number variants, and rare variants in protein coding genes will be determined by exome sequencing. The investigators will derive induced pluripotent stem cells from some participants to determine why CHD is so prevalent in TS. CHD risk genes will be identified in comparisons between TS cases with and without congenital heart defects. To facilitate these comparisons, the investigators will abstract the demographic and medical data of registry participants from questionnaires and medical records. Imaging will be used to confirm the diagnosis of CHD and to determine the prevalence and severity of additional cardiovascular defects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Turner Syndrome

Exclusion Criteria:

* Diagnosis excluding Turner Syndrome

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of females diagnosed with Turner Syndrome. This diagnosis can be based on physical symptoms (e.g. short stature, developmental delay, pubertal delay, etc.) or karyotype (e.g. 45X/46XX mosaic, 45X, etc.).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08-28 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Bicuspid aortic valve and thoracic aortic aneurysm | 10 years
  Imaging data

SECONDARY OUTCOMES:
Health-related quality of life | 10 years
  Access to care and guideline-recommended care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genetic and clinical IPD data will be shared with approved researchers with local IRB approval after authorization from the UTHouston study team. Aggregate data will be made available to the general research community through NIH databases.